CLINICAL TRIAL: NCT06840821
Title: A Phase I/II, Multicenter, Open-label, Single-arm, Dose-escalation and Dose-expansion Study Evaluating the Safety, Tolerability, and Preliminary Anti-tumor Activity of MB0151 Sequential Therapy in Adult Subjects With Advanced Solid Tumors (Including Gastroenteropancreatic Neuroendocrine Neoplasms, Small Cell Lung Cancer or Triple Negative Breast Cancer)
Brief Title: Evaluating the Safety, Tolerability, and Preliminary Anti-tumor Activity of MB0151 in Adult Subjects With Advanced Solid Tumors Expressing Somatostatin Receptors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mainline Biosciences (Shanghai) Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MB0151-101
Record Dates: First submitted 2025-02-07; First posted 2025-02-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MB0151 for injection (Experimental)
  Interventions: Drug: MB0151 for injection

INTERVENTIONS:
Drug: MB0151 for injection — In this study, the protocol of accelerated titration combined with i3+3 is used for dose escalation. administered intravenously every 2 weeks .

SUMMARY:
This is a multicenter, open-label, single-arm, dose-escalation and dose-expansion Phase I/II study to evaluate the safety, tolerability and preliminary anti-tumor activity of MB0151 in adult subjects (at least 18 years old) with advanced solid tumors. This study includes two phases: dose escalation and dose expansion. In this study, the protocol of accelerated titration combined with i3+3 is used for dose escalation,administered intravenously every 2 weeks. Enrolled subjects will be sequentially assigned to the planned dose cohorts according to this protocol to receive MB0151 treatment and will be monitored for the occurrence of DLT. The RP2D and/or OBD will be determined by considering the PK profile, safety and efficacy data in the dose-escalation stage (including backfill cohorts).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects over 18 years of age.
2. The subject must have a solid tumor confirmed by histology or cytology, and belong to one of the following categories: 1) locally advanced or metastatic SCLC, which has received standard treatment in the past and developed progress or intolerance; 2) Low-grade, medium-grade or high-grade locally advanced or metastatic GEP-NET, who has previously received first-line or multi-line anti-tumor treatment and developed progress or intolerance (unless there is no standard treatment available or such treatment is not suitable); 3) Metastatic or locally advanced unresectable TNBC, which is confirmed by histological examination, is characterized by the lack of expression of human epidermal growth factor 2(HER2), estrogen receptor (ER) and progesterone receptor (PR), and recurs/is refractory after standard treatment or has no standard treatment (which must include paclitaxel chemotherapy). 4) Other locally advanced or metastatic solid tumor subjects who have failed or are intolerant of standard treatment.
3. ECOG PS is 0-1.
4. Life expectancy ≥3 months.
5. Organ function is normal, which is defined as follows: 1) Bone marrow (not treated with blood transfusion or hematopoietic stimulating factors within 14 days): absolute neutrophil (ANC) ≥ 1.5× 10 9/L, platelet count ≥ 100× 10 9/L, hemoglobin ≥ 90 g/L. 2) Liver: total bilirubin (TBIL) ≤1.5× upper limit of normal value (ULN), or TBIL>1.5×ULN with direct bilirubin (DBIL) ≤ ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤3×ULN (≤5×ULN if accompanied by liver metastasis). 3) Kidney: serum creatinine concentration ≤1.5×ULN or creatinine clearance ≥50 mL/min(Cockcroft-Gault formula) 4) Coagulation function: partial thromboplastin activation time (APTT) or ≤ 1.5× ULN; International normalized ratio (INR) or prothrombin time (PT)≤1.5×ULN (INR<3.0 if the subject uses anticoagulant).
6. Detection requirements for biomarkers: 1) For the dose escalation and backfill cohort in Phase I study, biomarkers are not detected when they are selected, and the subjects need to provide archived or fresh tumor tissues within 2 years (if the archived tissue samples are more than 2 years and fresh tumor tissues are difficult to obtain, they can communicate with the applicant to decide whether to exempt them); During the study, the biomarker detection results of subjects in the follow-up dose expansion cohort may be added as additional selection criteria according to the obtained clinical data; 2) For Phase II study, the subjects should provide archived or fresh tumor tissues within 2 years (if the archived tissue samples are more than 2 years and fresh tumor tissues are difficult to obtain, they can communicate with the sponsor to decide whether to exempt them), and at baseline, the biomarkers should be detected by IHC in the central laboratory.
7. According to the RECIST version 1.1 standard, there is at least one target lesion (the target lesion must have not received radiotherapy before, or there is clear evidence of disease progression after radiotherapy).
8. Male or female subjects who are infertile, not in pregnancy or agree to use at least one effective contraceptive method during the study intervention period (from 14 days before the first administration to at least 180 days after the last administration of the study intervention) are eligible to participate in the study, and abide by the following contents: 1) Avoid donating fresh unwashed sperm or eggs. 2) Women who are breastfeeding should stop breastfeeding during the study period.
9. An informed consent form (ICF) that can be understood and signed, including compliance with ICF and the requirements and restrictions listed in this plan.

Exclusion Criteria:

1. According to the researcher's judgment, there are serious or poorly controlled systemic diseases, active bleeding tendency, renal transplantation or liver transplantation, active infection, including syphilis-specific antibody or human immunodeficiency virus (HIV) antibody positive, or active hepatitis B (hepatitis B surface antigen positive and/or core antibody positive and HBV-DNA copy number > 1000 copies /ml or > 200 IU/ml) or hepatitis C (C).
2. Suffering from other malignant tumors within 3 years before the first administration, except those who have received adequate treatment: 1) Cervical cancer in stage 1B or below. 2) Non-invasive basal cell or squamous cell skin cancer. 3) Non-invasive superficial bladder cancer. 4) Prostate cancer, the current PSA level is less than 0.1 ng/ mL.
3. Meet one or more of the following cardiac criteria: 1) Severe or unstable angina pectoris; 2) Myocardial infarction, coronary artery or peripheral artery bypass grafting, stroke or transient ischemic attack and symptomatic orthostatic hypotension occurred within 6 months before screening; 3) new york Heart Association II-IV heart failure; 4) QT interval (QTc) corrected by Fredericia formula at baseline: male > 450 msec, female > 470 msec；; 5) There are serious abnormalities in heart rhythm, conduction or morphology (for example, complete left bundle branch block, third degree heart block); 6) Congenital long QT syndrome; 7) Hypertension that is still poorly controlled after antihypertensive treatment (it needs to be measured three times continuously, that is, systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg).
4. Received major surgery within 28 days before C1D1.
5. There are unstable brain metastases with clinical symptoms and/or a history of meningeal diseases, brain stem or spinal cord compression. Subjects who have no clinical symptoms and have ≤3 metastatic lesions, and the largest lesion diameter is < <0.5cm, or whose symptoms are stable after treatment and do not need hormone drugs, can enter the study if they meet all the following criteria: (1) There are other measurable lesions besides the central nervous system; (2) New or expanded metastatic foci that have been in a stable state for at least 4 weeks without clinical evidence. If whole brain radiotherapy has been performed, it is at least 28 days before the first administration; If it is stereotactic radiosurgery or stereotactic radiotherapy, it is at least 14 days before the first administration.
6. Have a life-threatening trauma with increased risk of bleeding or a history of severe head trauma or intracranial surgery within 2 months before enrollment.
7. There is clear imaging evidence of tumor cavity or large blood vessel invasion, and the tumor is adjacent to important blood vessel structures, and the researcher judges that there is a risk of fatal bleeding.
8. Peripheral motor neuropathy or peripheral neuropathy with CTCAE grade ≥2 exists.
9. There are active viral, bacterial or fungal infections with clinical significance, which need the following treatment: 1) start intravenous antibacterial treatment within 4 weeks before the first administration, or 2) start oral antibacterial treatment within 10 days before the first administration.
10. Suffering from inflammatory bowel diseases, including Crohn's disease and ulcerative colitis.
11. Pneumonia ≥ 3 or clinically significant lung diseases, such as interstitial lung disease, non-infectious pneumonia, radiation pneumonia, pulmonary fibrosis, acute lung injury, etc.; Moderate and severe asthma and chronic obstructive pulmonary disease (COPD) requiring long-term drug treatment.

12 suffering from acute or chronic inflammatory skin diseases that have not yet recovered.

13. Have a history of deep venous thrombosis, pulmonary embolism or other serious venous thromboembolism within 3 months before the first administration (implantable venous access or catheter-derived thrombosis or superficial venous thrombosis is not considered as serious venous thromboembolism).

14. There is pelvic cavity, abdominal cavity, chest cavity or pericardial effusion that needs intervention, which can be included in the subjects in a stable state (the amount of effusion is not significantly increased and there are no clinical symptoms when the drainage tube is pulled out or undrained, and it lasts for at least 14 days).

15. The subject has a history of immunodeficiency diseases, including congenital and acquired immunodeficiency diseases.

16. Ophthalmology: There were active ocular surface diseases at baseline (based on ophthalmic evaluation). Have a history of cicatricial conjunctivitis (evaluated by an ophthalmologist). 1) There are active ocular surface diseases at baseline (based on ophthalmic evaluation). 2) Have a history of cicatricial conjunctivitis (evaluated by an ophthalmologist). Previous/combined treatment 17. Previous treatment distance before the first drug administration (C1D1): 1) Systemic anti-tumor treatment, including chemotherapy, biotherapy, immunotherapy, chemoembolization, or interventional chemotherapy, was received within 28 days or 5 half-lives (whichever is shorter). 2) receiving mitomycin C and nitrosourea drugs (such as carmustine [BiCNU or BCNU], lomustine, etc.) within 6 weeks; 3) Within 2 weeks or 5 half-lives (whichever is shorter), they have received oral fluorouracil (FU), small-molecule targeted antitumor drugs and endocrine therapy; 4) Received traditional Chinese medicine/Chinese patent medicine treatment with anti-tumor indications within 2 weeks; 5) receive radical radiotherapy within 4 weeks and palliative radiotherapy within 2 weeks; 6) Use powerful CYP3A inhibitors or inducers within 2 weeks or 5 half-lives (whichever is shorter).

18. Vaccinated with live attenuated vaccine within 4 weeks before the first administration of the study drug, or expected to need to be vaccinated with live attenuated vaccine during the study period.

19. Received corticosteroid (prednisone or equivalent dose of corticosteroid) with cumulative dose ≥150 mg within 2 weeks before the first infusion.

20. Previous treatments with coupled or uncoupled orestatin derivatives, including verbotezumab, verbotezumab, vintoizumab, vidiximab, vitexozumab, etc.

21. Any previous AE related to antineoplastic drugs must be restored to Grade ≤1, but it does not include alopecia, endocrine abnormality/vitiligo, or Grade 2 neurotoxicity caused by previous treatment (excluding peripheral and sensory neuropathy), unless the researcher thinks that these symptoms are not expected to cause excessive risk to the subjects or adversely affect their participation in this study.

22. Participate in other interventional clinical research at the same time, except for observational (non-interventional) research or in the follow-up period of interventional research.

23. Known past or current suffering from coagulation defects that increase the risk of bleeding.

24. Suffering from unhealed massive hemorrhage is defined as: 1) symptomatic hemorrhage of key regional organs, such as intracranial, intraocular, retroperitoneal, intra-articular or pericardial, or intramuscular hemorrhage with osteofascial compartment syndrome; 2) Hemorrhage occurred within 14 days before 2)C1D1, which led to a decrease in hemoglobin level of ≥20 g/L(0.31 mmol/L), or hemorrhage caused by transfusion of ≥2 units of whole blood or red blood cells.

25 allergic to octreotide or other somatostatin analogues or have a history of allergic reactions; Allergy to the study drug or payload or its derivatives or a history of immediate allergic reaction.

26. Other circumstances that the researcher thinks may cause excessive risks to the subjects, or may adversely affect their participation in this study, and the researcher judges that they are not suitable to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2028-07-04 (Estimated); Study Completion 2028-07-04 (Estimated)

PRIMARY OUTCOMES:
Phase I: Incidence of AEs, SAEs, infusion-related AEs, administration site AEs, AEs with CTCAE Grade ≥ 3 and AEs related to the investigational product | up to 2 years
Phase I: Incidence of DLT, MTD | From the first dose to 28 days
Phase I: ECG QTc Interval | up to 2 years
Phase I: OBD for dose-expansion study | up to 2 years
Phase II: ORR | up to 2 years
Phase II: DOR | up to 2 years
Phase II: DCR | up to 2 years
Phase II: PFS | up to 2 years
Phase II: OS | up to 2 years

SECONDARY OUTCOMES:
Phase I: Cmax | up to 2 years
Phase I:Tmax | up to 2 years
Phase I: AUC0-t | up to 2 years
Phase I: AUC0-∞ | up to 2 years
Phase I: t1/2 | up to 2 years
Phase I: CL | up to 2 years
Phase I: Vss | up to 2 years
Phase I: Incidence and severity of adverse events of interest | up to 2 years
  Phase I: Incidence and severity of adverse events of interest, including: MB0151-related peripheral neuropathy, hepatotoxicity, rash and skin reactions, infusion-related reactions, hemorrhage events, neutropenia, eye lesions, elevated blood glucose and diabetes mellitus
Phase I: Anti-drug antibody (ADA) positive rate | up to 2 years
Phase I: Objective Response Rate (ORR) | up to 2 years
Phase I: Duration of Response (DOR) | up to 2 years
Phase I: Disease Control Rate (DCR) | up to 2 years
Phase I: Progression-Free Survival (PFS) | up to 2 years
Phase I: Overall Survival (OS) | up to 2 years
Phase II: Incidence of AEs, SAEs, infusion-related AEs, administration site AEs, AEs with CTCAE Grade ≥ 3 and AEs related to the investigational product | up to 2 years
Phase II: Cmax | up to 2 years
Phase II: Cmin | up to 2 years
Phase II: ADA positive rate | up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Affiliated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No